CLINICAL TRIAL: NCT06401135
Title: Effects of Different Inspiratory Muscle Training Protocols on Functional Exercise Capacity and Respiratory and Peripheral Muscle Strength in Patients With Chronic Kidney Disease: A Randomized Study
Brief Title: Effects of Different Inspiratory Muscle Training Protocols in Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Nihan Katayıfçı, assistant professor, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hatay Mustafa Kemal U 2
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Chronic Kidney Diseases; Inspiratory Muscle Training; Exercise Capacity
Keywords: Chronic kidney disease; Inspiratory muscle training
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to the following groups: Group 1 (10% MIP), Group 2 (30% MIP), or Group 3 (60% MIP).
Who Masked: Participant
Masking Description: The patients will be not informed about their groups and they will be evaluated and trained at different places and times
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): Group 1 will receive inspiratory muscle training (IMT) using threshold loading device (POWERbreathe Classic, IMT Technologies Ltd. Birmingham, England) at 10% of maximal inspiratory pressure (MIP).
  The MIP will be measured at supervised session each week, and 10% of measured MIP value will be the new training workload.
  The treatment group will train for 30 min-per/day, 7 days/week, for 8 weeks. Six sessions at home and 1 session will be performed at department.
  Interventions: Other: Inspiratory muscle training
- Low intensity inspiratory muscle training group (Experimental): Group 2 will receive inspiratory muscle training (IMT) using threshold loading device (POWERbreathe Classic, IMT Technologies Ltd. Birmingham, England) at 30% of maximal inspiratory pressure (MIP).
  The MIP will be measured at supervised session each week, and 30% of measured MIP value will be the new training workload.
  The treatment group will train for 30 min-per/day, 7 days/week, for 8 weeks. Six sessions at home and 1 session will be performed at department.
  Interventions: Other: Inspiratory muscle training
- High intensity inspiratory muscle training group (Experimental): Group 3 will receive inspiratory muscle training (IMT) using threshold loading device (POWERbreathe Classic, IMT Technologies Ltd. Birmingham, England) at 60% of maximal inspiratory pressure (MIP).
  The MIP will be measured at supervised session each week, and 60% of measured MIP value will be the new training workload.
  The treatment group will train for 30 min-per/day, 7 days/week, for 8 weeks. Six sessions at home and 1 session will be performed at department.
  Interventions: Other: Inspiratory muscle training

INTERVENTIONS:
Other: Inspiratory muscle training — IMT will be conducted using a pressure threshold-loading device (POWERbreathe® Classic Low Resistance). The groups will train for 30 min-per/day, 7 days/week, for 8 weeks. Six sessions at home and 1 session will be performed at department. physiotherapist

SUMMARY:
The goal of this study is to investigate the effects of different IMT protocols on respiratory muscle strength, functional exercise capacity, quadriceps femoris muscle strength (QMS), handgrip muscle strength (HGS), QoL, respiratory function, dyspnoea, fatigue, balance, and PA levels in patients with CKD that were not on dialysis.

DETAILED DESCRIPTION:
Peripheral and respiratory muscle weakness has been reported in patients with chronic kidney disease (CKD). Management of respiratory muscle weakness is crucial, as reduced functional performance is related to respiratory muscle weakness.

Different IMT function protocols with 30-70% of the maximal inspiratory pressure (MIP) have been found to improve these in patients with CKD. The most efficient IMT intensity for patients with CKD is unknown. Therefore, this study aims to investigate the effects of different IMT protocols on respiratory muscle strength, functional exercise capacity, quadriceps femoris muscle strength (QMS), handgrip muscle strength (HGS), QoL, respiratory function, dyspnoea, fatigue, balance, and PA levels in patients with CKD that were not on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD stages 1-5 based on the CKD staging proposed by the Kidney Disease Outcomes Quality Initiative who are not on dialysis
* Aged>18 years
* No change in medications over one month

Exclusion Criteria:

* Uncontrolled hypertension
* Non-stable cardiac disease
* Recent viral infections
* Respiratory, neurological, and orthopedic diseases
* Pregnant and lactating patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscle strength | First day
  A mouth pressure device will be used to evaluate IMS.

SECONDARY OUTCOMES:
Functional exercise capacity | First day
  Functional exercise capacity will be evaluated with 6 minutes working test. Test will be performed in an enclosed 30-m corridor. The patients walk as fast as they could within 6 min.
Peripheral muscle strength | First day
  A hand-held dynamometer will be used to measure peripheral muscle strength. The measurements will be repeated three times, and the highest value will be used for comparison.
Expiratory muscle strength | First day
  A mouth pressure device will be used to evaluate EMS.
Pulmonary functions FEV1 | First day
  Spirometry will be used to assess pulmonary function.
Pulmonary functions FVC | First day
  Spirometry will be used to assess pulmonary function.
Pulmonary functions FEV1/FVC | First day
  Spirometry will be used to assess pulmonary function.
Pulmonary functions PEF | First day
  Spirometry will be used to assess pulmonary function.
Pulmonary functions FEF25-75% | First day
  Spirometry will be used to assess pulmonary function.
Dyspnoea | First day
  Dyspnoea will be measured using the Modified Medical Research Council (MMRC) dyspnoea scale. Levels of dyspnea are graded 0-4.
Fatigue | First day
  Fatigue will be assessed using the Fatigue Severity Scale (FSS). The total score ranges from 0 to 7.
Quality of life assessment | First day
  The Short Form 36 (SF-36) questionnaire will be used to assess QoL and includes both physical and mental components. The scores range from 0 to 100.
Physical activity | First day
  Physical activity will be assesed using the International Physical Activity Questionnaire (IPAQ) short form, which includes questions on sitting duration, walking activity, and moderate and vigorous activities.The IPAQ is categorized as inactive (<600 MET-min/week), minimally active (600-3000 MET-min/week), and sufficiently active (>3000 MET-min/week) based on total scores.
Balance | First day
  Balance will be evaluated using the Berg Balance Scale (BBS). The scale includes 14 items scoring 0 to 4. Higher scores indicate better balance.

CONTACTS AND LOCATIONS:
Overall Officials: Nihan Katayıfçı, Study Chair — Mustafa Kemal University
Locations (1):
- Hatay Mustafa Kemal University, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill NR, Fatoba ST, Oke JL, Hirst JA, O'Callaghan CA, Lasserson DS, Hobbs FD. Global Prevalence of Chronic Kidney Disease - A Systematic Review and Meta-Analysis. PLoS One. 2016 Jul 6;11(7):e0158765. doi: 10.1371/journal.pone.0158765. eCollection 2016. PMID 27383068
- [Background] de Lima MC, Cicotoste Cde L, Cardoso Kda S, Forgiarini LA Jr, Monteiro MB, Dias AS. Effect of exercise performed during hemodialysis: strength versus aerobic. Ren Fail. 2013;35(5):697-704. doi: 10.3109/0886022X.2013.780977. Epub 2013 Apr 8. PMID 23560491
- [Background] de Medeiros AIC, Fuzari HKB, Rattesa C, Brandao DC, de Melo Marinho PE. Inspiratory muscle training improves respiratory muscle strength, functional capacity and quality of life in patients with chronic kidney disease: a systematic review. J Physiother. 2017 Apr;63(2):76-83. doi: 10.1016/j.jphys.2017.02.016. Epub 2017 Mar 14. PMID 28433237
- [Background] Zhang F, Wang H, Bai Y, Huang L, Zhang H. Effect of respiratory muscle training in patients with chronic kidney disease: A systematic review and meta-analysis of randomized controlled trials. Clin Rehabil. 2023 Mar;37(3):348-361. doi: 10.1177/02692155221135729. Epub 2022 Nov 3. PMID 36325749
- [Derived] Katayifci N, Huzmeli I, Iri S D, Turgut FH. Effects of different inspiratory muscle training protocols on functional exercise capacity and respiratory and peripheral muscle strength in patients with chronic kidney disease: a randomized study. BMC Nephrol. 2024 May 29;25(1):184. doi: 10.1186/s12882-024-03610-1. PMID 38811888